CLINICAL TRIAL: NCT00530296
Title: Effectiveness of Cognitive Behavioral Therapy in Patients With End-Stage Renal Disease in Hemodialysis and With Depression
Brief Title: CBT to Treat Depression in Renal Patients
Acronym: CBTRPat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04/08710-8
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Depression; End Stage Renal Disease
Keywords: Depression; End stage renal disease; Quality of Life; Cognitive Behavioral Therapy
MeSH Terms: conditions — Depression; Kidney Failure, Chronic | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Group therapy, 12 sessions (90 minutes each, one session per week) manual "Coping with depression course"

SUMMARY:
The purpose of this study is to determine whether Cognitive Behavioral Therapy is effective in the treatment of depression in patients with end-stage renal disease in hemodialysis therapy

DETAILED DESCRIPTION:
Depression is a persistent problem among patients with end-stage renal disease and it does not tend to improve over time. The implementation of effective interventions to treat and prevent recurrence of depressive episodes is needed. The objectives of this study are: 1)the detection of Major Depression in hemodialysis patients; 2)to allocate patients with depression in two groups: structured program of treatment with CBT (group therapy)and control group (conventional psychotherapy at the dialysis unit); and 3)to verify whether after 3 months of CBT there was a remission of depressive symptoms and a improvement of the quality of life in the CBT group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Chronic renal disease (end stage) in hemodialysis for at least 3 months
* Diagnosis of Major depression disorder (4 or more clinical criteria in MINI and a BDI score of 10 or more)

Exclusion Criteria:

* Patients in process of renal transplant with (living donor)
* Psychiatric comorbidity
* Cognitive impairment or mental retardation
* Current substance abuse
* Heart failure, angina pectoris, arrhythmias

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-06; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Mini International Neuropsychiatric Interview (MINI-DSM-IV) Beck Depression Inventory (BDI) | Baseline; 3 months (end of intervention); follow-up (6 months after the end of the intervention)

SECONDARY OUTCOMES:
Kidney Disease and Quality of Life Short-form (KDQOL-SF) | Baseline; 3 months (end of intervention); follow-up (6 months after the end of the intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Priscila S. Duarte, MA, Principal Investigator — Federal University of Sao Paulo (UNIFESP); Ricardo CS Sesso, PhD, Study Chair — Federal University of Sao Paulo (UNIFESP); Maria Cristina OS Miyazaki, PhD, Study Chair — FAMERP Medical School
Locations (1):
- Priscila Silveira Duarte, São José do Rio Preto, São Paulo, Brazil